CLINICAL TRIAL: NCT02557282
Title: CARESTREAM Vue PACS v12.1.5 CT Perfusion Clinical Protocol
Acronym: CTP
Status: Completed | Type: Observational
Sponsor: Carestream Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 9J8421
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-03

CONDITIONS: Ischemia
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Predicate software: Olea Sphere PACS with CT Perfusion Module
- Investigational software: Vue PACS 12.1.5 Computed Tomography (CT) Perfusion

SUMMARY:
The purpose of this clinical study is to evaluate the CARESTREAM Vue PACS 12.1.5 Computed Tomography (CT) Perfusion ("investigational device") imaging performance. Evaluation of CT Perfusion (CTP) imaging will compare CTP with the predicate device, the Olea Sphere PACS with CT Perfusion Module.

DETAILED DESCRIPTION:
This study will demonstrate the imaging performance CTP by an assessment of 30 CTP de-identified patient cases collected retrospectively. The purpose of the study is to demonstrate equivalent clinical quality between the investigational and predicate devices using a radiologist evaluation of key metrics which are applicable to CTP images.

The maps include the following:

* Mean Transfer Time (MTT) - the time that the contrast material stays in the tissue
* Cerebral Blood Volume (CBV) - the volume of blood that is in a known volume of the tissue based on the concentration of contrast material that is in the tissue over the time
* Cerebral Blood Flow (CBF) - describes the flow of the blood to the affected tissue
* Time To Peak (TTP) - the time that maximum enhancement is achieved at each volume of the tissue
* Time to maximum of impulse response function (TMAX)

The retrospective data collected for each patient will include a non-contrast head CT exam completed on the same day as CTP image, and a follow-up head CT at least 1-2 days after the initial imaging study (initial non-contrast head CT) if available.

Similar performance between the investigational and predicate devices was demonstrated by the following criteria.

i. Substantial equivalence of the perfusion maps between devices ii. Substantial equivalence of the core and penumbra tissues resulting from thresholds on the perfusion maps between devices iii. The clinical decision based on the exclusion or inclusion criteria for treatment is equivalent between devices

ELIGIBILITY:
Inclusion Criteria:

* Retrospective patient CTP cases with case maps that include the following information: MTT, CBV, CBF, TTP, and TMAX.
* Initial CT exam and CT exam 1-2 days after the initial exam if available, and
* Retrospective CTP case with subject/patient 18 years of age or older

Exclusion Criteria:

* Low quality images, or images that are not clinically acceptable for clinical diagnostic reading as determined by the Principal Investigator,
* Subject less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty retrospective CT perfusion (CTP) cases that include the collection of CTP original data, perfusion maps and 2 non-contrast head CTs.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
To compare the diagnostic value of CTP in CARESTREAM Vue PACS ("investigational device") to the Olea Sphere PACS with CT Perfusion Module ("predicate device"). | one month
  Demonstrate equivalent clinical quality between the investigational and predicate devices.

CONTACTS AND LOCATIONS:
Overall Officials: Ayelet Eran, MD, Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: No